CLINICAL TRIAL: NCT00679094
Title: Phase I Single Dose Safety and Pharmacokinetic Study of a New Formulation of Bowman Birk Inhibitor Concentrate, Delivered as an Orange Juice Suspension to Healthy Male Volunteers Between 18 and 65 Years of Age
Brief Title: Bowman-Birk Inhibitor Concentrate in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00865; NCI-2009-00865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000595863; UPCC-N01-CN-25118-2; UPCC-805938; UPCC-805938 (Other: Abramson Cancer Center of The University of Pennsylvania); N01-CN-25118-2 (Other: DCP); P30CA016520 (NIH); N01CN25118 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy, no Evidence of Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm I (Experimental): Participants receive a single dose of oral BBIC or placebo, as an orange juice suspension, immediately followed by consumption of a defined low-fat breakfast. Participants continue to consume a low-fat diet for the next 48 hours and then resume their normal diet.
  Interventions: Drug: Bowman-Birk inhibitor concentrate; Other: placebo; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Bowman-Birk inhibitor concentrate — Given orally
  Other Names: BBIC
Other: placebo — Given orally
  Other Names: PLCB
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of Bowman-Birk inhibitor concentrate in healthy men. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of Bowman-Birk inhibitor concentrate may prevent cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the toxicity of single-dose Bowman-Birk Inhibitor Concentrate (BBIC) when administered as a suspension in orange juice in healthy male participants.

II. Determine the appropriate dose range and doses to be used in a subsequent phase I multiple-dose BBIC study that will be based upon the data gathered from this phase I single-dose study.

III. Characterize the pharmacokinetics of single-dose BBIC.

OUTLINE: This is a dose-escalation study of Bowman-Birk Inhibitor Concentrate (BBIC). Participants are sequentially assigned to 1 of 4 dose level cohorts. One participant in each dose level cohort is randomized to receive placebo or BBIC.

Participants receive a single dose of oral BBIC or placebo, as an orange juice suspension, immediately followed by consumption of a defined low-fat breakfast. Participants continue to consume a low-fat diet for the next 48 hours and then resume their normal diet.

Participants undergo blood and urine sample collection periodically for pharmacokinetic studies. Samples are analyzed by a sandwich enzyme-linked immunosorbent assay to measure concentrations of BBIC and its metabolites in serum and urine.

After completion of study treatment, participants are followed once weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participant recruited from the Philadelphia, Pennsylvania metropolitan area
* ECOG performance status 0-2
* WBC ≥ 3,000/uL
* Differential (i.e., neutrophils, lymphocytes, monocytes, bands, eosinophils, and basophils) normal
* Platelet count normal
* Hemoglobin normal
* Hematocrit normal
* RBC normal
* Creatinine normal
* Bilirubin normal
* ALT and AST normal
* Amylase and lipase normal
* Glucose normal
* Cholesterol normal
* Triglycerides normal
* Non-smoker

  * Former smokers are eligible provided they have not smoked within the past 3 months
* Within 15% of ideal body weight based on standard weight tables
* No vegetarians or individuals who normally ingest large amounts of soy products, defined as two or more servings of tofu, soy milk, or other primarily soy-based food per day
* No prior allergy or adverse reaction to soybeans
* No diagnosis of cancer within the past 5 years except nonmelanoma skin cancer
* No prior diagnosis of pancreatitis, pancreatic carcinoma, pancreatic adenoma, diabetes mellitus, obstruction of pancreatic ducts, or amyloidosis
* No history of heart disease
* EKG normal (normal variants allowed)
* No evidence of psychiatric problems
* No history of excessive alcohol consumption (i.e., an average of > 2 alcoholic beverages per day)
* No alcohol consumption within the past 3 days
* No history of any medical condition that could influence gastrointestinal uptake of the drug
* No history of chronic medical condition
* No evidence of another life-threatening disease
* More than 12 months since prior chemotherapy
* More than 1 month since prior experimental drugs
* More than 2 weeks since prior and no concurrent regular use (i.e., > 3 times/week) of nonsteroidal anti-inflammatory drugs (NSAIDs)
* More than 2 weeks since prior and no concurrent multivitamin tablets (or other vitamin supplements) of > 2 per day

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose, defined as the highest dose level at which none of the subjects in that dose group experience DLT as measured by NCI Common Toxicity Criteria | Up to 48 hours
Pharmacokinetics of BBIC in the serum as measured by a sandwich enzyme-linked immunosorbent assay | Immediately before BBIC administration and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 after administration
  Presented in a form of time course of serum BBI concentration after BBIC ingestion by the study subjects and peak concentration (Cmax), time to reach peak concentration (Tmax), area under the curve (AUC), and elimination rate constant (kel) and serum half-lives (t1/2) will be calculated for each subject. Mean, median, and 95% confidence interval will then be calculated for each parameter for each dose group. The relationship between dose and the above parameters will be investigated using simple linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States